CLINICAL TRIAL: NCT06599515
Title: A Multicenter Comparative Prospective Observational Cohort Study About Robot-assisted Laparoscopic Inguinal Hernia Repair Using Two Different Robotic Systems
Brief Title: SetUp Study for HugoTM RAS Inguinal Hernia Repair
Acronym: SUSHI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Filip Muysoms, Principal Investigator, Algemeen Ziekenhuis Maria Middelares
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUSHI
Record Dates: First submitted 2024-08-20; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Inguinal Hernia
Keywords: robot-assisted laparoscopic inguinal hernia repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: HugoTM Ras (Medtronic) robotic system
Masking Description: daVinci Xi (Intuitive Surgical) robotic system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HugoTM Ras (Medtronic) robotic system (Active Comparator): The patient is positioned supine position and a tilt of Trendelenburg of 12 degrees is given. A Verres needle insufflation at Palmers' point at the left subcostal margin will be done to achieve a pneumoperitoneum of 12 mmHg. Subsequently, a trocar of 12 mm is placed at the upper margin of the umbilicus using an optical trocar. Two further trocars of 8 mm are placed left and right side at 7 to 8 cm distance from the umbilical trocar and 2 cm caudal from the umbilical trocar. The setup of the arms, tilt and angles are done using the setup guide. The operation is performed using a scope with a 0°-degree angle. As instruments we have a fenestrated bipolar forceps in the left hand and a monopolar curved scissors in the right hand. Mesh used will be DextileTM Anatomical Mesh X-Large of 16x12 cm. There is a left sided and a right sided version and in bilateral hernias the meshes will overlap on the midline. The peritoneum is closed using a barbed suture (V-Loc 3/0) of 15 cm in length.
  Interventions: Procedure: robotic surgical platform
- daVinci Xi (Intuitive Surgical) robotic system (Active Comparator): An 8-mm trocar will be placed at the supraumbilical position after creation of pneumoperitoneum using a Verress needle with an intra-abdominal pressure of 12 mmHg. Two additional trocars (8 mm) are placed bilaterally in the flank at the level of the umbilicus under direct vision. The distance between the lateral trocars and the umbilical trocar will be 7 cm at minimum. The Progrip™ Laparoscopic Self-Fixating Mesh of 12×16 cm (anatomic version, Medtronic, Minneapolis, MN, US) will be used. The suture will be a slowly absorbable barbed suture 15 cm in length (V-Loc™ 90, Medtronic, Minneapolis, MN, US). The trocars are docked to the robotic arms, with the endoscope at the umbilicus. Inguinal hernia repair will be performed according to the standard surgical principle.
  Interventions: Procedure: robotic surgical platform

INTERVENTIONS:
Procedure: robotic surgical platform — robot-assisted laparoscopic inguinal hernia repair (rTAR)

SUMMARY:
The goal of this observational cohort study is to evaluate the evolution of the operative time in performing robotic assisted laparoscopic inguinal hernia repair (rTAPP) during the learning curve of the first 50 patients using the HugoTM Ras (Medtronic) robotic system using the setup guide.

Researchers will compare to the operative time for rTAPP of 50 patients by the same surgeon in another hospital using the daVinci Xi (Intuitive Surgical) robotic system.

DETAILED DESCRIPTION:
As a result of human cadaveric sessions to evaluate the approach of inguinal hernia repair using the Hugo RAS robotic system a setup guide was produced. Preclinic tests on dummies, cadaveric models and porcine models were performed. During a first session using dummies, the existing set-up guide proposed by US surgeons was tested and validated.

To evaluate the evolution of the operative time in performing robotic assisted laparoscopic inguinal hernia repair (rTAPP) during the learning curve of the first 50 patients using the HugoTM Ras (Medtronic) robotic system using the setup guide at the Sint Vincentius Hospital in Deinze. This will be compared to the operative time for rTAPP of 50 patients by the same surgeon in General hospital Maria Middelares using the daVinci Xi (Intuitive Surgical) robotic system.

Patient data and outcome data will be collected. A follow-up of 1 month postoperative is foreseen for the evaluation of short-term complications and quality of life 1 month after surgery.

ELIGIBILITY:
Inclusion Criteria: All patients planned for a minimal invasive (robotic assisted laparoscopic) inguinal hernia repair during the study period will be invited to take part in the study. Both unilateral and bilateral hernias will be included.

Exclusion Criteria:

* Recurrent hernias after previous preperitoneal mesh placement.
* Inguinal hernias after abdominal prostatectomy.
* Pregnancy.
* Emergency surgery.
* Age below 18 years.
* Absence of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Operative times | Minutes, up to 4 hours
  Comparison of operative times for rTAPP

SECONDARY OUTCOMES:
Short-term complications | until 30 days after the surgical procedure
  Evaluation of short term complications
Quality of Life (QoL) one month after surgery | until 30 days after the surgical procedure
  Evaluation of quality of life 1 month after surgery, using the EuraHS Quality of Life questionnaire, a lower score means a better quality of life

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - AZ Sint-Vincentius, Deinze
  - AZ Maria Middelares, Ghent

IPD SHARING:
Plan to Share IPD: No